CLINICAL TRIAL: NCT07348887
Title: Phase II Randomized Trial of RT-Led Daily Adaptive Radiotherapy for Submandibular Gland-Sparing in Head and Neck Cancer (RTL-DART)
Brief Title: Phase II Study of Daily Adaptive Radiotherapy for Submandibular Gland-sparing in Head and Neck Cancer
Acronym: RTL-DART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-5273
Record Dates: First submitted 2025-11-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Cancer of Head and Neck (SCCHN)
MeSH Terms: interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image guided radiation therapy (Active Comparator): This arm will proceed as per the standard of care. The pre-treatment reference plan will be delivered daily for 35 fractions. If a notable change in anatomy is identified, a dose of the day calculation may be performed as per current standard head and neck workflow
  Interventions: Radiation: Image guided radiation therapy
- Daily Adaptive Radiation Therapy (Experimental): Structures of daily adaptive radiation therapy organ at risk will be AI generated in the Ethos platform on the daily CBCT and then edited by radiation therapy team as required. A rigid registration of CTV targets to the CBCT replicating the current radiation therapy led IGRT process.
  Interventions: Radiation: Daily adaptive radiation therapy

INTERVENTIONS:
Radiation: Daily adaptive radiation therapy — Adaptive radiotherapy (ART) is the modification of the radiotherapy plan during treatment to account of changes from the original anatomy and set up. Reduction in treatment volume can be achieved through ART by:
  1. adjusting for gradual longitudinal changes in tumour and anatomy
  2. adjusting to account for uncertainty in set up and anatomy via daily online
  Other Names: Daily ART; DART
  Arms: Daily Adaptive Radiation Therapy
Radiation: Image guided radiation therapy — The pre-treatment reference plan will be delivered daily for 35 fractions.
  Other Names: IGRT
  Arms: Image guided radiation therapy

SUMMARY:
This is a randomized, single centre, single blinded prospective study comparing the standard of care imaging guided radiation therapy and daily adaptive radiotherapy (ART) for submandibular gland-sparing in head and neck cancer

DETAILED DESCRIPTION:
This study will recruit up to 50 patients planned to receive curative (chemo) radiotherapy for (head and neck squamous cell carcinoma) HNSCC with at least one level 1b lesion not being treated electively and with no high dose structure <1cm to spared (submandibular gland) SMG. The effect of daily ART with SMG dose sparing will be studied using both doimetric analysis and externally-validated quantitative metrics of unstimulated salivary flow as an object assessment for submandibular gland function. Patient report outcomes will assess the effect of the intervention on self-reported quality of life following treatment.

Patients, at the time of enrollment, will be randomized into one of the two treatment arms. The patients will be blinded to prevent bias in their quality of life assessments.

Patients in both arms will undergo a baseline functional CT scan along with other assessments including oral and dental assessment, PSS-HNC swallow assessment, unstimulated salivary flow rate test, DMFS160 index, and quality of life questionnaire. The radiation treatment will take approximately 7 weeks to complete. The follow up visits will be at 1.5, 6, 12, and 24 months with assessments similar to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically proven Squamous Cell carcinoma of head and neck
* Bilateral neck being treated
* At least one level 1b not being treated electively and with no target structure, other than elective level II/III, <1cm to spared SMG
* ECOG PS 0-2
* Planned for curative (chemo)radiotherapy
* Able to receive and understand verbal and written information regarding study and able to give written informed consent
* Be able to lie comfortably on back and to wear immobilization for up to 1 hour

Exclusion Criteria:

* As judged by investigator evidence of systemic disease that makes unsuitable for study
* Pregnancy
* Underlying salivary dysfunction prior to treatment judged by investigator to affect likelihood of benefit from ART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in saliva production | 6 months
  Change in saliva production from baseline measured by MST (Malnutrition Screening Test) at 6 months following IGRT or daily ART HN treatment

SECONDARY OUTCOMES:
Change in saliva production | 24 months
  Saliva production measured by MST (Malnutrition Screening Test) during radiotherapy and at 1.5, 12 and 24 months
MDADI (MD Anderson Dysphagia Inventory) | 24 months
  Patient reported outcomes at baseline, end of treatment and 1.5, 6, 12 and 24 months. Low score means low functioning. High score means high functioning/healthy.
Swallow assessment | 24 months
  Swallow assessment via performance status scale (PSS) for Head and Neck Cancer (PSS-HNC) at baseline, end of treatment and 1.5, 6, 12 and 24 months. Higher score means high functional/healthy.
Toxicity assessment | 24 months
  Clinician assessed toxicity at baseline, weekly during radiotherapy and 1.5, 6, 12,and 24 months (CTCAE v5). Low grade side toxicity and less number of toxicities means patients are healthier compared to high grade and high number of toxicities.
Comparing dental health between two arms | 24 months
  Dental health following treatment (Dental assessment + DMFS 160 index). DMFS stands for Decayed, Missing, Filled Surfaces. Low score means healthy teeth and gums.
Procedure delivery comparison | 24 months
  Analysis of average time and staff requirements to deliver daily ART versus IGRT
Xerostomia questionnaire | 24 months
  Patient reported qualitative measurements at baseline, end of treatment and 1.5, 6, 12 and 24 months. Lower score means that patients are producing an adequate amount of saliva. High score means their mouths are dry.
EORTC QLQ HN43 (Quality of Life Questionnaire Head and Neck 43) | 24 months
  Patient reported qualitative measurements at baseline, end of treatment and 1.5, 6, 12 and 24 months. Low score means that patients do not have problems in their daily life. High score means they are having more difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada